CLINICAL TRIAL: NCT01424631
Title: Single Incision Versus Conventional Laparoscopic Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel-Raouf El-Geidie, assistant professor general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: lap appendectomy 123
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- single incision laparoscopic appendectomy (Active Comparator)
  Interventions: Procedure: single incision laparoscopic appendectomy
- conventional laparoscopic appendectomy (Placebo Comparator)
  Interventions: Procedure: conventional laparoscopic appendectomy

INTERVENTIONS:
Procedure: single incision laparoscopic appendectomy
  Arms: single incision laparoscopic appendectomy
Procedure: conventional laparoscopic appendectomy
  Arms: conventional laparoscopic appendectomy

SUMMARY:
This is a randomized prospective study comparing single incision versus conventional laparoscopic appendectomy for management of acute appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* acute appendicitis

Exclusion Criteria:

* perforation with peritonitis
* lower abdominal scar
* contraindications to laparoscopy

Ages: 10 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)